CLINICAL TRIAL: NCT03137901
Title: Agreement and Precision of Capstesia, a New Smarphone Application for PPV and CO Monitoring.
Acronym: Capstesia
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Other Study IDs: P2017/224 / B406201731906
Record Dates: First submitted 2017-04-19; First posted 2017-05-03 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Capstesia — Picture of the arterial waveform taken with a smartphone

SUMMARY:
This study test the agreement and precision of Pulse Pressure Variation (PPV) and Cardiac Output (CO) obtained by the Android application Capstesia™ against another pulse contour CO monitoring ( EV-1000, Edwards Lefesciences, USA)

DETAILED DESCRIPTION:
Pulse pressure variation (PPV) remains a good predictor of fluid responsiveness in the OR. However, PPV can be time-consuming to calculate (manual determination), is not always displayed on monitoring screens nor reliable through visual assessment and needs additional devices to be displayed. A new Android application (Captesia) automatically calculates the PPV utilizing a digital photograph of the arterial waveform from the monitor. The application determines the PPV by selecting peaks and troughs of the arterial curve.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for major surgery which requires a CO and PPV monitoring as standard of care

Exclusion Criteria:

* patients with arrhythmias like atrial fibrillation
* patients with valvular insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for major surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Agreement and precision of PPV and CO during 5 surgical phases (postinduction, pre incision, postincision, end of surgery and at least one episode of hypotension) | during surgery
  We will compare PPV and CO given with the EV-1000 and the capstesia app at different phases of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, M.D, Principal Investigator — Erasme
Locations (1):
- Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Joosten A, Jacobs A, Desebbe O, Vincent JL, Sarah S, Rinehart J, Van Obbergh L, Hapfelmeier A, Saugel B. Monitoring of pulse pressure variation using a new smartphone application (Capstesia) versus stroke volume variation using an uncalibrated pulse wave analysis monitor: a clinical decision making study during major abdominal surgery. J Clin Monit Comput. 2019 Oct;33(5):787-793. doi: 10.1007/s10877-018-00241-4. Epub 2019 Jan 3. PMID 30607806